CLINICAL TRIAL: NCT03797898
Title: Well-Child Care Clinical Practice Redesign: A Parent Coach-Led Model of Care for Young Children
Brief Title: Well-Child Care Clinical Practice Redesign: A Parent Coach-Led Model of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tumaini Coker, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000413; 5R01HD088586 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2019-01-09 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Preventive Health Services; Health Promotion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents will meet with a Parent Coach during child's routine well visits, and have access to the parent coach between visits for additional follow up and concerns, and have access to a preventive care text messaging services (Healthy Txt).
  Interventions: Other: Parent Coach
- Control (No Intervention): usual care well child care

INTERVENTIONS:
Other: Parent Coach — The Parent Coach intervention uses a health educator who provides anticipatory guidance, psychosocial screening/ referral, and developmental/behavioral surveillance, screening, and guidance at each well-visit. The Parent Coach uses a parent-focused, pre-visit questionnaire to customize the visit to the parents' needs. Every well-visit includes a brief, problem-focused encounter with a clinician for a physical exam and any concerns that require a clinician's attention. Finally, an automated text message service provides for periodic, age-specific messages to reinforce key health messages from Parent Coach-led well-visits.
  Arms: Intervention

SUMMARY:
Parent-focused Redesign for Encounters, Newborns to Toddlers (PARENT) is a team-based approach to care using a health educator ("Parent Coach") to provide the bulk of WCC services, address specific needs faced by families in low-income communities, and decrease reliance on the clinician as the primary provider of WCC services. The Parent Coach provides anticipatory guidance, psychosocial and social needs screening/referral, and developmental and behavioral surveillance, screening, and guidance at each WCC visit, and is supported by parent-focused pre-visit screening and visit prioritization, a brief, problem-focused clinician encounter for a physical exam and any concerns that require a clinician's attention, and an automated text message parent reminder and education service for periodic, age-specific messages to reinforce key health-related information recommended by Bright Futures national guidelines.

The investigators will conduct a cluster RCT of PARENT to determine its effects on quality, utilization, and clinician efficiency, and its cost/cost-offset.

DETAILED DESCRIPTION:
Well-Child Care (WCC) visits for child preventive care during the first three years of life are critical because they may be the only opportunity before a child reaches preschool to identify and address important social, developmental, behavioral, and health issues that could have significant impact and long-lasting effects on children's lives as adults. Despite its potential, multiple studies have demonstrated that pediatric providers fail to provide all recommended preventive and developmental services at these visits and that most parents leave the visit with unaddressed psychosocial, developmental, and behavioral concerns. Further, these missed opportunities are more pronounced for children in low-income families.

A critical problem is that the structure of WCC in the U.S. cannot support the vast array of WCC needs of families. Key structural problems include (a) reliance on clinicians (pediatricians, family physicians, or nurse practitioners) for basic, routine WCC services, (b) limitation to a 15-minute face-to-face clinician-directed WCC visit for the wide array of education and guidance services in WCC, and (c) lack of a systematic, patient-driven method for visit customization to meet families' needs. These structural problems contribute to the wide variations in processes of care and preventive care outcomes, resulting in poorer quality of WCC and perhaps worse health outcomes, particularly for children in low-income communities.

To address the gaps in current WCC this study introduces a new model of care to meet the needs of children in low-income communities: Parent-focused Redesign for Encounters, Newborns to Toddlers (PARENT). PARENT is a team-based approach to care using a health educator ("Parent Coach") to provide the bulk of WCC services, address specific needs faced by families in low-income communities, and decrease reliance on the clinician as the primary provider of WCC services. The Parent Coach provides anticipatory guidance, psychosocial screening/referral, and developmental and behavioral surveillance, screening, and guidance at each WCC visit, and is supported by parent-focused pre-visit screening and visit prioritization, a brief, problem-focused clinician encounter for a physical exam and any concerns that require a clinician's attention, and an automated text message parent reminder and education service for periodic, age-specific messages to reinforce key health-related information recommended by Bright Futures national guidelines.

To assess the efficacy of PARENT, the investigators will conduct a cluster randomized controlled trial (RCT). The study will be conducted in partnership with 10 clinics.

In preparation for the trial, investigators will use a Community Engagement & Intervention Implementation process that has been successful in previous studies to guide the intervention adaptation process, Parent Coach training, practice workflow, and intervention implementation in the practices. For the study trial, the investigators will conduct a cluster RCT of PARENT to determine its effects on quality, utilization, and clinician efficiency, and its cost/cost-offset. The project's community partners include two federally-qualified health centers (FQHC). FQHC #1 has 4 clinics participating in the study and FQHC #2 has 6 clinics participating in the study. The total number of clinics participating in the study is 10 clinics randomized at the clinic level to intervention or control condition. The intervention clinics will implement PARENT for all well-visits through age 2 years at their clinical site, and the control clinics will continue usual care (clinician directed well-visit). 1,000 families will be enrolled at infant age ≤12 months and remain in the study for a period of 12 months. Parents will complete a survey at baseline and at 6 and 12-months post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian-Child dyad attending well child check-up visits for a 2-week to 12- month WCC visit.
* Parent is English or Spanish proficient
* For multiple gestations, one infant will be randomly selected as the index child. Infants with special health care needs will not be excluded from the study, since these children generally need the same recommended preventive care services.

Exclusion Criteria:

* More than one child attending Well-Child Care
* Legal guardian of child is under 18 years of age
* Parents who are employed by one of the federally-qualified health centers (FQHCs)
* Parents/legal guardian not planning to continue receiving well child care services at this clinic for their child in the next 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 937 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tumaini R Coker, MD/MBA, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mimila NA, Chung PJ, Elliott MN, Bethell CD, Chacon S, Biely C, Contreras S, Chavis T, Bruno Y, Moss T, Coker TR. Well-Child Care Redesign: A Mixed Methods Analysis of Parent Experiences in the PARENT Trial. Acad Pediatr. 2017 Sep-Oct;17(7):747-754. doi: 10.1016/j.acap.2017.02.004. Epub 2017 Feb 14. PMID 28232142
- [Background] Coker TR, Chacon S, Elliott MN, Bruno Y, Chavis T, Biely C, Bethell CD, Contreras S, Mimila NA, Mercado J, Chung PJ. A Parent Coach Model for Well-Child Care Among Low-Income Children: A Randomized Controlled Trial. Pediatrics. 2016 Mar;137(3):e20153013. doi: 10.1542/peds.2015-3013. Epub 2016 Feb 10. PMID 26908675
- [Background] Coker TR, Windon A, Moreno C, Schuster MA, Chung PJ. Well-child care clinical practice redesign for young children: a systematic review of strategies and tools. Pediatrics. 2013 Mar;131 Suppl 1(Suppl 1):S5-25. doi: 10.1542/peds.2012-1427c. PMID 23457149
- [Background] Coker TR, Moreno C, Shekelle PG, Schuster MA, Chung PJ. Well-child care clinical practice redesign for serving low-income children. Pediatrics. 2014 Jul;134(1):e229-39. doi: 10.1542/peds.2013-3775. Epub 2014 Jun 16. PMID 24936004
- [Derived] Coker TR, Lowry SJ, Dwibedi E, Salaguinto T, Szilagyi PG, Fiscella K, Rangel SJ, Ortiz J, Weaver MR. Cost Analysis of the PARENT Trial of Community Health Workers in Early Childhood Preventive Care: A Secondary Analysis of a Cluster-Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2522732. doi: 10.1001/jamanetworkopen.2025.22732. PMID 40742591
- [Derived] Coker TR, Liljenquist K, Lowry SJ, Fiscella K, Weaver MR, Ortiz J, LaFontaine R, Silva J, Salaguinto T, Johnson G, Friesema L, Porras-Javier L, Guerra LJS, Szilagyi PG. Community Health Workers in Early Childhood Well-Child Care for Medicaid-Insured Children: A Randomized Clinical Trial. JAMA. 2023 May 23;329(20):1757-1767. doi: 10.1001/jama.2023.7197. PMID 37120800
- [Derived] Hurst R, Liljenquist K, Lowry SJ, Szilagyi PG, Fiscella KA, Weaver MR, Porras-Javier L, Ortiz J, Sotelo Guerra LJ, Coker TR. A Parent Coach-Led Model of Well-Child Care for Young Children in Low-Income Communities: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 25;10(11):e27054. doi: 10.2196/27054. PMID 34842563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two multi-site federally qualified health centers (FQHCs) in California and Washington State, with 6 and 4 participating practices each. The first participant was enrolled March 5, 2019 and the last participant was enrolled July 1, 2021. **PLEASE NOTE that there were not multiple phases to the trial. this study was a cluster RCT that did not have multiple phases to the trial.
Pre-assignment Details: Of 937 enrolled participants, 914 remained enrolled and were eligible to complete 12-month follow-up.
  Participants are unique parent/child dyads. The parents were enrolled and each parent had an index child that they provided data on. This was the child for who they were coming to the clinic for a well child visit, and the child had to be 12 months of age or younger.
Units Other Than Participants: clinics
Groups:
- Intervention: Clinics assigned to the intervention arm will use the Parent Coach model for well child care visits, for children ages 0-2. Parents will meet with a Parent Coach during child's routine well visits, and have access to the parent coach between visits for additional follow up and concerns, and have access to a preventive care text messaging services (Healthy Txt).
  Parent Coach: The Parent Coach intervention uses a health educator who provides anticipatory guidance, psychosocial screening/ referral, and developmental/behavioral surveillance, screening, and guidance at each well-visit. The Parent Coach uses a parent-focused, pre-visit questionnaire to customize the visit to the parents' needs. Every well-visit includes a brief, problem-focused encounter with a clinician for a physical exam and any concerns that require a clinician's attention. Finally, an automated text message service provides for periodic, age-specific messages to reinforce key health messages from Parent Coach-led well-visits.
- Control: Clinics assigned to control group use usual well child care. They do not have a parent coach as part of the visit.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 452; 5 clinics (452 parent participants with a child ≤12 months arriving for a well child visit) | 485; 5 clinics (485 parent participants with a child ≤12 months arriving for a well child visit)
Completed | 378; 5 clinics | 407; 5 clinics
Not Completed | 74; 0 clinics | 78; 0 clinics
Not completed — Lost to Follow-up | 60 | 69
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Became ineligible | 5 | 2

BASELINE CHARACTERISTICS:
Population: participants are parent/child dyads. Each dyad includes 1 parent with 1 child. there is no overlap-- so that the number of parents is equal to the number of children in the study. each parent/child dyad is from a unique family. This is the overall number of participants (914) contributing baseline data. Not all participants answered every baseline question, so the number for each of the baseline measures does not match with the total participating.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 438 | 476 | 914
Age, Continuous [Mean (Standard Deviation); unit: months] — Child Age (months). Parents reported on age of child. We did not collect data on parent age Population: 911 participants responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  months
    number analyzed (Participants) | 435 | 476 | 911
    (all) | 4.0 (4.0) | 4.7 (4.0) | 4.4 (4.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participant (parent/caregiver) relationship to child. Child sex/gender was not collected. Population: 911 respondents responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    Mother: number analyzed (Participants) | 435 | 476 | 911
    Mother | 414 | 454 | 868
    Father: number analyzed (Participants) | 435 | 476 | 911
    Father | 20 | 22 | 42
    Grandmother: number analyzed (Participants) | 435 | 476 | 911
    Grandmother | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants] — Parent race/ethnicity (child race/ethnicity not collected) Population: 911 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  participants
    Latino: number analyzed (Participants) | 437 | 474 | 911
    Latino | 321 | 343 | 664
    Non-Latino Black: number analyzed (Participants) | 437 | 474 | 911
    Non-Latino Black | 24 | 22 | 46
    Non-Latino Asian: number analyzed (Participants) | 437 | 474 | 911
    Non-Latino Asian | 14 | 13 | 27
    Non-Latino White: number analyzed (Participants) | 437 | 474 | 911
    Non-Latino White | 52 | 56 | 108
    Non-Latino Multi-Racial: number analyzed (Participants) | 437 | 474 | 911
    Non-Latino Multi-Racial | 16 | 15 | 31
    Non-Latino Other: number analyzed (Participants) | 437 | 474 | 911
    Non-Latino Other | 10 | 25 | 35
Primary language spoken at home [Count of Participants; unit: Participants] — Parent reported parent primary language spoken at home Population: 913 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 437 | 476 | 913
    English | 212 | 243 | 455
    Spanish | 197 | 199 | 396
    Other | 28 | 34 | 62
Respondent country of birth [Count of Participants; unit: Participants] — Parent reported parent country of birth Population: 912 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 436 | 476 | 912
    United States | 218 | 249 | 467
    Country other than U.S. | 218 | 227 | 445
Respondent marital status [Count of Participants; unit: Participants] — Parent reported parent marital status Population: 913 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 437 | 476 | 913
    Married | 164 | 181 | 345
    Divorced | 6 | 8 | 14
    Living with a partner | 165 | 189 | 354
    Separated | 13 | 12 | 25
    Single (never married & currently not living with a partner) | 89 | 86 | 175
Number of adults in the home [Count of Participants; unit: Participants] — Population: 913 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 437 | 476 | 913
    1 adult | 21 | 23 | 44
    2 adults | 232 | 257 | 489
    3 adults | 67 | 82 | 149
    4 or more adults | 117 | 114 | 231
Number of children that parent has [Count of Participants; unit: Participants] — Population: 913 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 437 | 476 | 913
    1 child | 144 | 169 | 313
    2 children | 130 | 126 | 256
    3 children | 82 | 105 | 187
    4 or more children | 81 | 76 | 157
Child health insurance [Count of Participants; unit: Participants] — Parent reported insurance type for enrolled child Population: 912 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 436 | 476 | 912
    Medicaid (Medi-Cal/Apple Health) | 405 | 450 | 855
    Private Insurance Plan | 7 | 7 | 14
    Military | 1 | 0 | 1
    Uninsured | 17 | 15 | 32
    More than one | 4 | 3 | 7
    Unknown | 2 | 1 | 3
Child chronic medical problems [Count of Participants; unit: Participants] — Parent report of enrolled child chronic medical problems Population: 912 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 436 | 476 | 912
    Chronic medical problems | 10 | 6 | 16
    No chronic medical problems | 426 | 470 | 896
Trouble paying for any household expenses [Count of Participants; unit: Participants] — Parent report of "some" or "a lot" of trouble paying for any household expenses in the past 12 months Population: 907 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 432 | 475 | 907
    Trouble paying for any household expenses in past 12 months | 238 | 289 | 527
    No trouble paying for any household expenses in past 12 months | 194 | 186 | 380
Highest level of education completed [Count of Participants; unit: Participants] — Parent highest level of education Population: 912 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 436 | 476 | 912
    Less than high school | 111 | 120 | 231
    High school graduate or GED | 159 | 166 | 325
    2-Year college or some college | 127 | 152 | 279
    4-Year college degree or greater | 39 | 38 | 77
Household Annual Income [Count of Participants; unit: Participants] — Parent reported household annual income Population: 768 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 370 | 398 | 768
    < $29,999 per year | 246 | 236 | 482
    $30,000 to $49,999 per year | 83 | 111 | 194
    $50,000 to $69,999 per year | 25 | 29 | 54
    $70,000 or more | 16 | 22 | 38
Child's current overall health [Count of Participants; unit: Participants] — Parent reported child's current overall health Population: 908 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  Participants
    number analyzed (Participants) | 433 | 475 | 908
    Excellent | 293 | 325 | 618
    Very good | 89 | 105 | 194
    Good | 43 | 44 | 87
    Fair/poor | 8 | 1 | 9
PROMIS (Patient-Reported Outcomes Measurement Information System) 2-item Global Mental Health [Mean (Standard Deviation); unit: T-Score] — PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population. PROMIS Mental Health was calculated by summing two 5-point Likert scale questions for a total possible of 2-10 (9 values), then converting those sums to corresponding PROMIS T-scores, for 9 T-score values ranging from 25.8-64.6. Higher scores represent better outcomes. https://staging.healthmeasures.net/images/PROMIS/manuals Population: 906 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  T-Score
    number analyzed (Participants) | 432 | 474 | 906
    (all) | 54.7 (8.5) | 53.9 (8.2) | 54.3 (8.3)
PROMIS (Patient-Reported Outcomes Measurement Information System) 2-item Global Physical Health [Mean (Standard Deviation); unit: T-Score] — PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population. PROMIS Physical Health was calculated by summing 2 5-point Likert scale questions for a total possible of 2-10 (9 values), then converting those sums to corresponding PROMIS T-scores, for 9 T-score values ranging from 23.4-63.3. Higher scores represent better outcomes. https://staging.healthmeasures.net/images/PROMIS/manuals Population: 907 respondents of 914 responded to this item.Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  T-Score
    number analyzed (Participants) | 432 | 475 | 907
    (all) | 51.1 (8.4) | 50.6 (7.9) | 50.9 (8.2)
PROMIS (Patient-Reported Outcomes Measurement Information System) 4-item Emotional Support Score [Mean (Standard Deviation); unit: T-Score] — PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population. PROMIS Emotional Support was calculated by summing 4 5-point Likert scale questions for a total possible of 4-20 (17 values), then converting those sums to corresponding PROMIS T-scores, for T-score values ranging from 25.7-62.0. Higher scores represent better outcomes. https://staging.healthmeasures.net/images/PROMIS/manuals Population: 905 respondents of 914 responded to this item. Number analyzed differs from overall because of missing data (participant did not respond to item in question)
  T-Score
    number analyzed (Participants) | 430 | 475 | 905
    (all) | 57.6 (7.0) | 57.2 (7.6) | 57.4 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Preventive Care Services: Anticipatory Guidance Topics Received by Parent Report at Well Visits
Description: Using anticipatory guidance items adapted from the Promoting Healthy Development Survey, the investigators will assess whether parents receive the recommended anticipatory guidance topics.
  scale, 0-100, higher is better
Time Frame: 12 months post enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 375 | 407
score on a scale | 73.9 (23.4) | 63.3 (27.8)

2. Primary Outcome: Healthcare Utilization: Emergency Department Utilization
Description: any emergency department care visit for the index child in past 12 months (parent report)
Time Frame: 12 months post enrollment
Population: all participants completing 12 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 376 | 407
Participants | 140 | 147

3. Secondary Outcome: Clinician Time With Parent During the Well-Child Care (WCC) Visit, From Observations of Well Child Care Visit
Description: time spent in parent-provider visit during the well child care visit. these data were not collected for trial participants at baseline. At follow-up, we did not collect data due to pandemic restrictions in doing observations.
Time Frame: Data not collected due to COVID Pandemic restrictions on in clinic observations.
Population: Data were not collected due to COVID 19 pandemic restrictions on in clinic observations
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Receipt of Preventive Care Services: Psychosocial Screening Received by Parent Report at Well Visits
Description: Using items adapted from the Promoting Healthy Development Survey, the investigators will assess whether parents received psychosocial assessment on all 7 items
Time Frame: 12 months post enrollment
Population: all participants completing 12 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 407
Participants | 253 | 203

5. Secondary Outcome: Receipt of Preventive Care Services: Developmental Concerns Addressed and Screening Received by Parent Report at Well Visits.
Description: Using items adapted from the Promoting Healthy Development Survey, the investigators will assess whether parents receive the recommended developmental screening and were asked if they had their developmental concerns addressed.
Time Frame: 12 months post enrollment
Population: Number analyzed differs from overall because of missing data (participant did not respond to item in question)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 407
Participants
  Behavioral Concerns Elicited & Addressed: number analyzed (Participants) | 342 | 356
  Behavioral Concerns Elicited & Addressed | 305 | 292
  Developmental Screening: number analyzed (Participants) | 363 | 394
  Developmental Screening | 310 | 332

6. Secondary Outcome: Healthcare Utilization: Hospitalizations
Description: any hospitalizations for index child in past 12 months by parent report
Time Frame: 12 months post enrollment
Population: all participants completing 12 month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 376 | 406
Participants | 12 | 9

7. Secondary Outcome: Healthcare Utilization: Well Child Care Visits Up to Date
Description: up to date on well child care by clinic electronic medical record review at 12 months post enrollment
Time Frame: 12 months post enrollment
Population: all enrolled participants who remained eligible, and consented to chart review by the 12-month post intervention assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 419 | 465
Participants | 309 | 295

8. Secondary Outcome: Experiences of Care: Helpfulness of Care Assessment by Parent Report
Description: parent reported helpfulness of care, using items adapted from Promoting Healthy Development Survey scale is 0-100, higher is better
Time Frame: 12 months post enrollment
Population: all participants completing 12 month survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 407
score on a scale | 77.8 (25.2) | 69.8 (30.7)

9. Secondary Outcome: Experiences of Care: Family Centeredness of Care- Whether it Was Received by Parent Report
Description: receipt of family centeredness of care using items adapted from National Survey of Children's Health scale 0-100, higher is better
Time Frame: 12 months post enrollment
Population: all participants completing 12 month survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 407
score on a scale | 89.0 (22.5) | 85.5 (27.1)

ADVERSE EVENTS:
Time Frame: 12 months
Description: As there were no risk of harm to participant dyads, we did not conduct a systematic approach to collecting data on harms. However, if in the course of the 12-month data collection, we gained information on participant harm to either the parent or child of the dyad, we report those as "adverse events". The only such information we received was on one parent of the parent/child dyads enrolled, and this event (parent death) is reported both in the serious adverse event and in all cause mortality.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/452 | 1/485
Serious Adverse Events (participants affected / at risk) | 0/452 | 1/485
Other Adverse Events (participants affected / at risk) | 0/452 | 0/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=452) | Control (N=485)
death (General disorders) | 0 (0) | 1 (1) — the parent enrolled in the study passed away during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03797898/Prot_SAP_000.pdf